CLINICAL TRIAL: NCT03768947
Title: Heat Therapy for Fibromyalgia: The Effect on Chronic Pain and Possible Mechanisms
Brief Title: Heat Therapy for Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Andrea Chadwick, MD, MSc, FASA, Assistant Professor, University of Kansas Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00142795
Record Dates: First submitted 2018-11-08; First posted 2018-12-07 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Fibromyalgia
Keywords: Chronic Pain
MeSH Terms: conditions — Fibromyalgia; Chronic Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Heat Therapy Arm (Experimental): Participants in this open-label pilot study will undergo heat therapy via hot water immersion (hot-tub).
  Interventions: Other: Heat therapy via hot water immersion

INTERVENTIONS:
Other: Heat therapy via hot water immersion — Participants will be asked to participate in a 4-week heat therapy intervention, which consists of ~12-15 visits (45 min each) of immersion in to a hot tub.

SUMMARY:
The purpose of this study is to see if heat therapy intervention via hot water immersion (i.e., a hot tub) is an effective treatment for patients with Fibromyalgia.

DETAILED DESCRIPTION:
Fibromyalgia (FM) is a complex and difficult-to-treat painful medical condition and is marked by chronic widespread musculoskeletal pain, decreased pain threshold, and comorbid symptomatology (e.g. fatigue, trouble thinking). Several factors appear to play a role in the pathophysiology of FM: abnormal pain processing, abnormal autonomic nervous and neuroendocrine system function, genetics, and environmental triggers. The prognosis for recovery in traditional medicine is generally poor and current pharmacological treatments for FM are often insufficient to control persistent symptoms. As such, complementary medicine and alternative lifestyle approaches are needed. Heat therapy, such as saunas and hot tubs, has been used historically for its presumed therapeutic benefits, and emerging research highlights the benefits of heat therapy on metabolic and cardiovascular disease risks. Finnish saunas, which result in total-body heating, have shown beneficial clinical effects for rheumatic patients and new studies are needed to determine if heat therapy could improve pain symptoms in patients with FM.

The short-term goal of the investigators is to determine, in a pilot clinical study, that heat therapy intervention via hot water immersion is a safe and efficacious treatment for pain in patients with FM. The overall hypothesis is that heat therapy intervention will improve clinical pain severity and associated dysfunction in a cohort of FM patients and that the anti-inflammatory actions of heat shock proteins may mediate this improvement. The proposed interdisciplinary study will provide data regarding treatment efficacy and will explore potential molecular and physiologic processes that may underlie improvement in pain symptoms after heat therapy intervention for FM. Furthermore, these key pilot studies will provide important preliminary data for future studies.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent provided by the participant
* Age 18 to 65 years
* Diagnosis of FM according to American College of Rheumatology 2011 self-report criteria64
* Average BPI visual numerical pain score > 4
* Stable doses of medications for at least 30 days prior to screening
* Participant agrees to continue the same medication regimen for the study duration
* FM patients with a sedentary lifestyle (exercise can alter heat shock protein levels)

Exclusion Criteria:

* Inability to provide informed consent
* Age greater than 65 years
* Previous history of hypotension
* Pregnancy
* Current clinically significant disease that would prevent safe heat therapy/hot water immersion (heart conditions such as myocardial infarction, angina, uncontrolled hypertension or kidney disease see below)
* Reported previous bleeding problems
* Anti-platelet medication (Plavix), Warfarin, and other anticoagulants (Eliquis, Pradaxa, and Xarelto)
* Recent rectal, anal, vaginal or prostate surgery
* Current litigation for fibromyalgia
* Current disability proceedings
* Active psychotic or suicidal symptoms
* Current drug or alcohol abuse
* Current regular exercise

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-07-19 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Visual Numerical Pain Score (VNS) at 1 month | Baseline and 1 Month
  Measured by the Brief Pain Inventory (BPI). The BPI scores are a numerical rating scale and range from 0 to 10. A score of 0 is equal to no pain and a score of 10 is equal to pain as bad as you can imagine.

SECONDARY OUTCOMES:
Change from Baseline Patient-Reported Outcomes Measurement Information System (PROMIS) at 1 month | Baseline to 1 Month
  PROMIS (Patient-Reported Outcomes Measurement Information System) measures to be included are Depression, Anxiety, Physical Functioning, and Sleep Impairment. Each questionnaire usually has 4-16 response options ranging in value from one to five. The total raw score for a short form with all questions answered is the sum of the values of the response to each question. The total range of potential raw scores depends on the number of questions being asked, for example, a 6 item form would have a range from is 6 to 30. After the raw score is calculated, a T-score metric is used to convert the raw score to a T-score. On the T-score metric, a score of 50 is the mean of a relevant reference population and 10 is the standard deviation of that mean. For PROMIS measures, higher scores equals "more of the concept being measured", this could be a desirable or undesirable outcome, depending on the concept being measured.
Change from Baseline Revised Fibromyalgia Impact Questionnaire (FIQ-R) at 1 month | Baseline and 1 Month
  The Revised Fibromyalgia Impact Questionnaire (FIQ-R) is a measure of symptom severity in fibromyalgia. There is a total of 21 questions and a range of scores from 0 to 210. The higher the score the more severe a person's symptoms.

OTHER OUTCOMES:
Quantitative Sensory Testing (QST)-- Pressure pain sensitivity by Multimodal Automated Sensory Testing | Baseline and 1 Month
  Pressure pain sensitivity is measured by the Multimodal Automated Sensory Testing (MAST) System (measured at the thumbnail). It yields a pressure pain threshold value measured in kg/cm2.
Blood Analyses of Change in Baseline Heat Shock Proteins at 1 month | Baseline and 1 Month
  Heat shock proteins including Heat Shock Protein 72 (HSP72), Heat Shock Factor 25 (HSP25), and Heat Shock Factor 1 (HSF1) will be measured via Western blots and Elisa assays in serum at baseline (pre-intervention) and post-intervention (within 48 hours of completion of the one month heat therapy intervention). Each of these specific heat shock proteins is measured as a protein to total protein ratio. For example, HSP25 is measured as HSP25/total protein.
Blood Analyses of Change in Pro/Anti-inflammatory Markers at 1 month | Baseline and 1 Month
  Pro/Anti-Inflammatory markers (IL-1Ra, IL-1β, IL-6, IL-8, IL-10, IL-18, IFN-α, TNF-α) will be measured via Western blots and Elisa assays in serum at baseline (pre-intervention) and post-intervention (within 48 hours of completion of the protocol). All markers will be measured as concentrations (nanograms/milliliter (ng/mL))

CONTACTS AND LOCATIONS:
Overall Officials: Andrea L Nicol, MD, Principal Investigator — University of Kansas School of Medicine; Paige Geiger, PhD, Principal Investigator — University of Kansas School of Medicine
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wolfe F, Clauw DJ, Fitzcharles MA, Goldenberg DL, Hauser W, Katz RS, Mease P, Russell AS, Russell IJ, Winfield JB. Fibromyalgia criteria and severity scales for clinical and epidemiological studies: a modification of the ACR Preliminary Diagnostic Criteria for Fibromyalgia. J Rheumatol. 2011 Jun;38(6):1113-22. doi: 10.3899/jrheum.100594. Epub 2011 Feb 1. PMID 21285161